CLINICAL TRIAL: NCT01528046
Title: A Phase I Trial of Dose Escalation of Metformin in Combination With Vincristine, Irinotecan, and Temozolomide in Children With Relapsed or Refractory Solid Tumors
Brief Title: Metformin in Children With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16962; SP003 (Other Grant/Funding Number: Pediatric Cancer Foundation)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumors; Primary Brain Tumors
Keywords: central nervous system (CNS); malignancy; relapsed; refractory; pediatric; recurrent
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Recurrence | interventions — Vincristine; Irinotecan; Temozolomide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin in Combination with VIT (Experimental): Participants will receive metformin in combination with vincristine, irinotecan and temozolomide (VIT).
  Interventions: Drug: Vincristine; Drug: Irinotecan; Drug: Temozolomide; Drug: Metformin

INTERVENTIONS:
Drug: Vincristine — Vincristine (VCR) = 1.5 mg/m^2/day (maximum dose 2 mg), days 1 and 8, administered as intravenous (IV) bolus over 1-5 minutes
  Other Names: VCR; Oncovin; NSC #067574; Vincristine sulfate
Drug: Irinotecan — Irinotecan (IRN) = 50 mg/m^2/day, days 1-5, IV over 60 minutes
  Other Names: CPT-11; Camptothecin-11; Camptosar ®; NSC#616348; IRN
Drug: Temozolomide — Temozolomide (TEM) = 50 mg/m^2/day by mouth (PO) Days 1-5
  Other Names: Temodar™; NSC #362856; TEM
Drug: Metformin — Metformin (MET) = dose as per dose escalation, divided twice a day (BID), PO continuously for the 21 day cycle.
  Other Names: Glucophage ®; MET

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of escalating doses of metformin on a backbone of vincristine, irinotecan and temozolomide (VIT) in children with recurrent and refractory solid tumors.

DETAILED DESCRIPTION:
Metformin is an oral anti-diabetes medication that activates AMP-activated protein kinase (AMPK). Recent data from in vitro and in vivo experiments, as well as epidemiologic retrospective analyses, suggest that metformin has anti-cancer activity. Vincristine, irinotecan, and temozolomide (VIT) is a combination of chemotherapeutic agents that have different mechanisms of action as well as disparate side effect profiles. Two recent phase 1 trials have demonstrated that this regimen is safe and well-tolerated in children with relapsed and refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be > 1 year of age and ≤ 18 years of age at time of initiation of protocol therapy.
* Diagnosis: Patients have a histologically or radiographically confirmed relapsed or refractory solid tumor or primary central nervous system (CNS) malignancy.
* Disease Status: Patients must have radiographically measurable disease.
* Therapeutic Options: Patients must have relapsed or refractory cancers for which there is no known curative option or other available therapy proven to prolong survival with an acceptable quality of life.
* Performance Level: Karnofsky ≥ 50% for patients older than 16 years old, and Lansky ≥ 50 for patients 1-16 years old.
* Prior Therapy: Patients may have received prior therapy including vincristine, irinotecan, or temozolomide. Patients may not have previously been treated with combination therapy of irinotecan and temozolomide.
* Patients must be fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  * Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of starting protocol therapy, or a minimum of six weeks must have elapsed since prior nitrosurea chemotherapy.
  * Hematopoietic growth factor: At least 7 days must have elapsed since the last administration of filgrastim, or 14 days since administration of pegfilgrastim.
  * Biologic (anti-neoplastic agent): At least 7 must have elapsed since the last administration of any biologic agent.
  * Radiation therapy (XRT): At least 14 days since the last dose of local palliative radiation therapy. Greater than 6 months must have elapsed since the last day of treatment if given total body irradiation, craniospinal irradiation.
  * Autologous or Allogenic Stem Cell Transplant: Complete resolution of graft versus host disease and no current need for immunosuppressive medication. Greater than 3 months must have elapsed since engraftment and no longer requiring transfusion of platelets or injection of colony stimulating factors.
* Organ Function Requirements

  * Bone Marrow Function: Peripheral absolute neutrophil count (ANC) ≥ 1000/μL; Platelet count ≥ 100,000/μL (no platelet transfusion within 7 days prior to obtaining laboratory result); Hemoglobin ≥ 8.0 gm/dL
  * Adequate Renal Function: Creatinine clearance or glomerular filtration rate ≥ 70ml/min/1.73m^2
  * Adequate Liver Function: Total bilirubin ≤ 1.5x upper limit of normal (ULN) for age; alanine transaminase (ALT) ≤ 5x ULN; Serum albumin ≥ 2gm/dL
* Informed Consent: All patients ≥ 18 years of age must sign a written informed consent. For patients < 18 years old, the patient's parents or legal guardians must sign a written informed consent, unless the patient is an emancipated minor. Childhood Assent, when age appropriate as per institutional guidelines, should be signed by the participating patient.

Exclusion Criteria:

* Significant organ dysfunction, not meeting inclusion criteria.
* Pregnancy or Breast-Feeding woman will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
* Concomitant Medications:

  * Growth factor: Growth factors that support platelet or white cell number of function must not have been administered within the past 7 days.
  * Steroids: Patients with CNS tumors who have not been on a stable or decreasing dose of dexamethasone for the past 7 days.
  * Investigational Drugs: Patients who are currently receiving another investigational drug.
  * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents.
  * Medication Allergy: Allergy or intolerance to agents on this protocol: vincristine, irinotecan, temozolomide, or metformin; Allergy to cephalosporins.
  * Infection: Patients who have uncontrolled infection, positive blood cultures within the past 48 hours, or receiving treatment for Clostridium difficile infection.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Average of 3 Months
  To determine the maximum tolerated dose (MTD) of metformin when given in conjunction with VIT in children with refractory and relapsed solid tumors.

SECONDARY OUTCOMES:
Number of Participants with Antitumor Activity | Average of 3 Months
  To evaluate the antitumor activity of the addition of metformin to VIT.
Pharmacokinetics | Average of 3 Months
  To describe the pharmacokinetics of metformin in children with relapsed malignancies receiving VIT combination chemotherapy.
Pharmacodynamics | Average of 3 Months
  To define the pharmacodynamics of metformin.
Metformin Concentrations | Average of 3 Months
  To determine tissue and tumor metformin concentrations in patients undergoing resection.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gill, M.D., Study Chair — The Children's Hospital at Montefiore, Pediatric Cancer Foundation, Sunshine Project; Damon Reed, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (14):
- United States (14):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Delaware, Wilmington, Delaware
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Children's Hospital at Montefiore, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Medical Center/Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Metts JL, Trucco M, Weiser DA, Thompson P, Sandler E, Smith T, Crimella J, Sansil S, Thapa R, Fridley BL, Llosa N, Badgett T, Gorlick R, Reed D, Gill J. A phase I trial of metformin in combination with vincristine, irinotecan, and temozolomide in children with relapsed or refractory solid and central nervous system tumors: A report from the national pediatric cancer foundation. Cancer Med. 2023 Feb;12(4):4270-4281. doi: 10.1002/cam4.5297. Epub 2022 Sep 23. PMID 36151773